CLINICAL TRIAL: NCT05453474
Title: Cell-based Non-invasive Prenatal Testing - Evaluation of Time of Blood Sampling and Whole Genome Amplification Prior to Genetic Testing
Brief Title: Cell-based Non-invasive Prenatal Testing as an Alternative to Invasive Chorionic Villus Sampling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Arcedi Biotech (Industry); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Christian Liebst Frisk Toft, Principal investigator, Molecular Biologist, ph.d., Aalborg University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: N-20180001 (cbNIPT v2)
Record Dates: First submitted 2022-02-17; First posted 2022-07-12 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Hereditary Diseases
Keywords: cell-based non-invasive prenatal testing; Hereditary disorders
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Intervention Model Description: All patients had either one or two blood samples collected. Each blood sampled had either all cells lyzed or cells were split between lysis and whole genome amplification. Hence, the study is considered to have to seperate analysis each with two arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WGA (Experimental): DNA from the cells are amplified by whole genome amplification prior to genetic testing.
  Interventions: Genetic: Whole genome amplification
- No-WGA (No Intervention): DNA from the cells are tested directly without whole genome amplification

INTERVENTIONS:
Genetic: Whole genome amplification — DNA is amplified by whole genome amplification
  Arms: WGA

SUMMARY:
The study aims to evaluate cell-based non-invasive prenatal testing (cbNIPT) as an alternative to invasive chorionic villus sampling (CVS) in patients who achieve pregnancy following preimplantation genetic testing for hereditary disorders.

DETAILED DESCRIPTION:
The study has three main objects:

1. to evaluate the optimal time of blood sampling (gestational week 7-8 or 11-14)
2. to evaluate whole genome amplification prior to genetic analysis og isolated fetal cells (only relevant for monogenic disorders)
3. evaluating specificity and sensitivity

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy following preimplantation genetic testing

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-08-08 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Evaluation of the fetal cell yield when blood sampling is performed at Gestational weeks 7-8 compared to gestational weeks 11-14. | Within 2 years
  Evaluation of whether cbNIPT be performed in gestational week 7-8.
Percentage of test with an informative test result from genetic testing following whole genome amplification or direct testing without whole genome amplification. | Within 2 years (since data analysis is carried out later than sample collection)
  Analysis of whether genetic testing on whole genome amplified material is inferior to genetic testing directly on DNA purified from single cells.
Specificity and sensitivity of single cell analysis. | Within 2 years
  Evaluation of the sensitivity and specificity of single cell analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Fertility Unit, Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Toft CLF, Ingerslev HJ, Kesmodel US, Hatt L, Singh R, Ravn K, Nicolaisen BH, Christensen IB, Kolvraa M, Jeppesen LD, Schelde P, Vogel I, Uldbjerg N, Farlie R, Sommer S, Ostergard MLV, Jensen AN, Mogensen H, Kjartansdottir KR, Degn B, Okkels H, Ernst A, Pedersen IS. Cell-based non-invasive prenatal testing for monogenic disorders: confirmation of unaffected fetuses following preimplantation genetic testing. J Assist Reprod Genet. 2021 Aug;38(8):1959-1970. doi: 10.1007/s10815-021-02104-5. Epub 2021 Mar 7. PMID 33677749
- See also: ARCEDI Biotech homepage — https://arcedi.com/